CLINICAL TRIAL: NCT03941873
Title: A Phase 1/2 Study to Investigate the Safety, Tolerability, Pharmacokinetics, and Preliminary Antitumor Activity of Sitravatinib as Monotherapy and in Combination With Tislelizumab in Patients With Unresectable Locally Advanced or Metastatic Hepatocellular Carcinoma or Gastric/Gastroesophageal Junction Cancer
Brief Title: A Study to Investigate Sitravatinib as Monotherapy and in Combination With Tislelizumab in Participants With Unresectable Locally Advanced or Metastatic Hepatocellular Carcinoma or Gastric/Gastroesophageal Junction Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BGB-900-104; CTR20182149 (Other: ChinaDrugTrials)
Record Dates: First submitted 2018-12-23; First posted 2019-05-08 (Actual); Results first posted 2024-10-18 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Carcinoma, Hepatocellular; Gastric/Gastroesophageal Junction Cancer
Keywords: Carcinoma; HCC; G/GEJ Cancer
MeSH Terms: conditions — Carcinoma, Hepatocellular; Carcinoma | interventions — sitravatinib; tislelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Sitravatinib Monotherapy: 80 mg (Experimental): Sitravatinib 80 mg orally once daily in 21-day cycles in participants with unresectable locally advanced or metastatic HCC or G/GEJ cancer
  Interventions: Drug: Sitravatinib
- Sitravatinib Monotherapy: 120 mg (Experimental): Sitravatinib 120 mg orally once daily in 21-day cycles in participants with unresectable locally advanced or metastatic HCC or G/GEJ cancer
  Interventions: Drug: Sitravatinib
- Sitravatinib 80 mg + Tislelizumab (Experimental): Sitravatinib 80 mg orally once daily in 21-day cycles with tislelizumab 200 mg intravenously (IV) once every 3 weeks in participants with unresectable locally advanced or metastatic HCC or G/GEJ cancer
  Interventions: Drug: Sitravatinib; Drug: Tislelizumab
- Sitravatinib 120 mg + Tislelizumab (Experimental): Sitravatinib 120 mg orally once daily in 21-day cycles with tislelizumab 200 mg IV once every 3 weeks in participants with unresectable locally advanced or metastatic HCC or G/GEJ cancer
  Interventions: Drug: Sitravatinib; Drug: Tislelizumab

INTERVENTIONS:
Drug: Sitravatinib — Administered orally as a capsule
  Other Names: MGCD516
Drug: Tislelizumab — Administered intravenously
  Other Names: BGB-A317; Tevimbra
  Arms: Sitravatinib 120 mg + Tislelizumab; Sitravatinib 80 mg + Tislelizumab

SUMMARY:
The purpose of this study was to evaluate the safety, tolerability, pharmacokinetics and preliminary antitumor activity of sitravatinib as monotherapy and in combination with tislelizumab in participants with unresectable locally advanced or metastatic hepatocellular carcinoma (HCC) or gastric/gastroesophageal junction (G/GEJ) cancer.

DETAILED DESCRIPTION:
This was an open-label, multicenter Phase 1/2 clinical study for participants with histologically or cytologically confirmed unresectable locally advanced or metastatic HCC or G/GEJ cancer. All participants received study treatment (s) until progressive disease, unacceptable toxicity, death, withdrawal of consent, or study termination by sponsor.

ELIGIBILITY:
Key Inclusion Criteria:

* Histologically or cytologically confirmed, unresectable, locally advanced, or metastatic HCC/gastric cancer/GEJ cancer
* Able to provide written informed consent and can understand and agree to comply with the requirements of the study and the schedule of assessments
* Age ≥ 18 years on the day of signing the informed consent form (or the legal age of consent in the jurisdiction in which the study is taking place)
* Adequate organ function
* Females of childbearing potential must be willing to use a highly effective method of birth control for the duration of the study, and ≥ 120 days after the last dose of study drug(s), and have a negative serum pregnancy test ≤ 7 days of first dose of study drug(s)
* Nonsterile males must be willing to use a highly effective method of birth control for the duration of the study and for ≥ 120 days after the last dose of study drug(s)
* Failed current standard-of-care treatment, or standard-of-care treatment is considered not appropriate at present

Key Exclusion Criteria:

* Active leptomeningeal disease or uncontrolled brain metastasis
* Active autoimmune diseases or history of autoimmune diseases that may relapse
* Any active malignancy ≤ 2 years before first dose of study drug(s)
* History of interstitial lung disease, noninfectious pneumonitis or uncontrolled diseases including pulmonary fibrosis or acute lung diseases
* Severe chronic or active infections (including tuberculosis infection) requiring systemic antibacterial, antifungal, or antiviral therapy within 14 days prior to first dose of study drug(s)
* Known history of human immunodeficiency virus (HIV) infection
* Untreated chronic hepatitis B or chronic hepatitis B virus (HBV) carriers.
* Any major surgical procedure requiring general anesthesia ≤ 28 days before the first dose of study drug(s)
* Prior allogeneic stem cell transplantation or organ transplantation
* Inadequately controlled hypertension (defined as systolic blood pressure > 150 mmHg and/or diastolic blood pressure > 100 mmHg)
* Bleeding or thrombotic disorders or use of anticoagulants such as warfarin or similar agents requiring therapeutic international normalized ratio (INR) monitoring
* Any systemic chemotherapy within 28 days of the first dose of study drug(s) or hormone therapy, targeted therapy, or any investigational therapies
* Toxicities (as a result of prior anticancer therapy) that have not recovered to baseline or stabilized, except for adverse events not considered a likely safety risk (eg, alopecia, neuropathy, and specific laboratory abnormalities)
* Inability to swallow capsules or disease significantly affecting gastrointestinal function
* Pregnant or breastfeeding woman

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2019-02-28 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — BeiGene
Locations (18):
- China (18):
  - The Second Hospital of Anhui Medical University, Hefei, Anhui
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Sun Yat Sen Memorial Hospital, Sun Yat Sen University (North), Guangzhou, Guangdong
  - Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Union Hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Zhongnan Hospital of Wuhan University Wuhan, Wuhan, Hubei
  - Hubei Cancer Hospital, Wuhan, Hubei
  - General Hospital of Eastern Theatre Command Qihuaiyuan Branch(the St Hospital of Chinese Pla), Nanjing, Jiangsu
  - The First Affiliated Hospital of Nanchang University Branch Donghu, Nanchang, Jiangxi
  - Liaoning Cancer Hospital and Institute, Shenyang, Liaoning
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Affiliated Zhongshan Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Shanghai East Hospital Branch Hospital, Shanghai, Shanghai Municipality
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Zhang, F., et al. Safety, tolerability, and preliminary antitumor activity of sitravatinib plus tislelizumab (TIS) in patients (pts) with unresectable locally advanced or metastatic hepatocellular carcinoma (HCC). Journal of Clinical Oncology 2022 40:4_suppl, 418; Meeting Abstract, 2022 ASCO Gastrointestinal Cancers Symposium; https://doi.org/10.1200/JCO.2022.40.4_suppl.418
- [Result] Chen Z., et al. Safety, tolerability, and preliminary antitumor activity of sitravatinib plus tislelizumab (TIS) in patients (pts) with unresectable locally advanced or metastatic gastric cancer/gastroesophageal junction cancer (GC/GEJC). Journal of Clinical Oncology 2022 40:4_suppl, 281-281; Meeting Abstract, ASCO Gastrointestinal Cancers Symposium, Abstract 281.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at multiple sites in China.
Groups:
- Sitravatinib Monotherapy: 80 mg: Sitravatinib 80 milligrams (mg) orally once daily in 21-day cycles in participants with unresectable locally advanced or metastatic hepatocellular carcinoma (HCC) or gastric/gastroesophageal junction (G/GEJ) cancer
Period: Overall Study
Arm/Group | Sitravatinib Monotherapy: 80 mg | Sitravatinib Monotherapy: 120 mg | Sitravatinib 80 mg + Tislelizumab | Sitravatinib 120 mg + Tislelizumab
Started | 3 | 24 | 3 | 81
Completed | 1 | 3 | 1 | 8
Not Completed | 2 | 21 | 2 | 73
Not completed — Death | 0 | 12 | 2 | 53
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 5
Not completed — Lost to Follow-up | 1 | 2 | 0 | 0
Not completed — Sponsor Decision | 0 | 6 | 0 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sitravatinib Monotherapy: 80 mg | Sitravatinib Monotherapy: 120 mg | Sitravatinib 80 mg + Tislelizumab | Sitravatinib 120 mg + Tislelizumab | Total
Number analyzed (Participants) | 3 | 24 | 3 | 81 | 111
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.7 (10.02) | 53.3 (9.92) | 56.3 (6.51) | 56.4 (10.23) | 55.7 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 1 | 10 | 14
  Male | 2 | 22 | 2 | 71 | 97
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian: Chinese | 3 | 24 | 3 | 81 | 111

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: Number of participants with treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs) per National Cancer Institute Common Terminology Criteria for Adverse Events Version 5.0 (NCI-CTCAE v5.0), including relevant physical examination, electrocardiograms, and laboratory assessments. Safety analysis set is presented by dose, as prespecified in the statistical analysis plan (SAP).
Time Frame: Up to approximately 4 years and 1 month
Population: The Safety Analysis Set includes all participants who received ≥ 1 dose of any study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Sitravatinib Monotherapy: 80 mg | Sitravatinib Monotherapy: 120 mg | Sitravatinib 80 mg + Tislelizumab | Sitravatinib 120 mg + Tislelizumab
Number analyzed (Participants) | 3 | 24 | 3 | 81
Participants
  At least one TEAE | 3 | 24 | 3 | 78
  At least one SAE | 1 | 7 | 2 | 31

2. Primary Outcome: Objective Response Rate (ORR)
Description: ORR is defined as the percentage of participants whose best overall response (BOR) is the confirmed complete response (CR) or partial response (PR) assessed by investigator using Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. Efficacy evaluable analysis set is presented by indication group, as prespecified in the statistical analysis plan.
Time Frame: Up to approximately 4 years and 1 month
Population: The Efficacy Evaluable Analysis Set includes all participants who received ≥ 1 dose of any study drug with measurable disease at baseline per RECIST v1.1 and who had ≥ 1 evaluable postbaseline tumor assessment unless treatment was discontinued due to clinical progression or early death (within 13 weeks after the first dose date) before tumor assessment
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Sitravatinib Monotherapy: Sitravatinib 80 mg or 120 mg orally once daily in 21-day cycles in participants with anti-programmed cell death protein-1 and anti-PD ligand-1 (PD-1/PD-L1) antibody naïve or refractory/resistant (R/R) HCC
- Sitravatinib + Tislelizumab: Sitravatinib 80 mg or 120 mg orally once daily in 21-day cycles with tislelizumab 200 mg IV once every 3 weeks in participants with anti-PD-1/PD-L1 antibody naïve or R/R HCC and anti-PD-1/PD-L1 antibody naïve G/GEJ cancer
Arm/Group | Sitravatinib Monotherapy | Sitravatinib + Tislelizumab
Number analyzed (Participants) | 20 | 78
Percentage of participants
  Anti-PD-1/PD-L1 naïve or R/R HCC: number analyzed (Participants) | 20 | 0
  Anti-PD-1/PD-L1 naïve or R/R HCC | 25.0 [8.7 to 49.1] |
  Anti-PD-1/PD-L1 naïve HCC: number analyzed (Participants) | 0 | 26
  Anti-PD-1/PD-L1 naïve HCC |  | 11.5 [2.4 to 30.2]
  Anti-PD-1/PD-L1 R/R HCC: number analyzed (Participants) | 0 | 21
  Anti-PD-1/PD-L1 R/R HCC |  | 9.5 [1.2 to 30.4]
  Anti-PD-1/PD-L1 naïve G/GEJ cancer: number analyzed (Participants) | 0 | 31
  Anti-PD-1/PD-L1 naïve G/GEJ cancer |  | 16.1 [5.5 to 33.7]

3. Secondary Outcome: Duration of Response (DOR)
Description: DOR is defined as the time from the first determination of an objective response until the first documentation of progressive disease as assessed by investigator per RECIST v1.1, or death, whichever comes first. Results are reported for indication groups with responders, defined as complete response (CR) or partial response (PR). Efficacy evaluable analysis set is presented by indication group, as prespecified in the statistical analysis plan.
Time Frame: Up to approximately 4 years and 1 month
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Sitravatinib Monotherapy: Sitravatinib 80 mg or 120 mg orally once daily in 21-day cycles in participants with anti-PD-1/PD-L1 antibody naïve or R/R HCC
Arm/Group | Sitravatinib Monotherapy | Sitravatinib + Tislelizumab
Number analyzed (Participants) | 5 | 10
Months
  Anti-PD-1/PD-L1 naïve or R/R HCC: number analyzed (Participants) | 5 | 0
  Anti-PD-1/PD-L1 naïve or R/R HCC | 7.7 [2.8 to NA] — NA = not estimable due to low number of participants with events |
  Anti-PD-1/PD-L1 naïve HCC: number analyzed (Participants) | 0 | 3
  Anti-PD-1/PD-L1 naïve HCC |  | 5.7 [4.1 to NA] — NA = not estimable due to low number of participants with events
  Anti-PD-1/PD-L1 R/R HCC: number analyzed (Participants) | 0 | 2
  Anti-PD-1/PD-L1 R/R HCC |  | NA [5.4 to NA] — NA = not estimable due to low number of participants with events
  Anti-PD-1/PD-L1 naïve G/GEJ cancer: number analyzed (Participants) | 0 | 5
  Anti-PD-1/PD-L1 naïve G/GEJ cancer |  | 5.5 [2.7 to NA] — NA = not estimable due to low number of participants with events

4. Secondary Outcome: Disease Control Rate (DCR)
Description: DCR is defined as the percentage of participants with BOR as CR, PR, or stable disease (SD) assessed by investigator per RECIST v1.1. Efficacy evaluable analysis set is presented by indication group, as prespecified in the statistical analysis plan.
Time Frame: Up to approximately 4 years and 1 month
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Sitravatinib Monotherapy | Sitravatinib + Tislelizumab
Number analyzed (Participants) | 20 | 78
Percentage of participants
  Anti-PD-1/PD-L1 naïve or R/R HCC: number analyzed (Participants) | 20 | 0
  Anti-PD-1/PD-L1 naïve or R/R HCC | 90.0 [68.3 to 98.8] |
  Anti-PD-1/PD-L1 naïve HCC: number analyzed (Participants) | 0 | 26
  Anti-PD-1/PD-L1 naïve HCC |  | 84.6 [65.1 to 95.6]
  Anti-PD-1/PD-L1 R/R HCC: number analyzed (Participants) | 0 | 21
  Anti-PD-1/PD-L1 R/R HCC |  | 81.0 [58.1 to 94.6]
  Anti-PD-1/PD-L1 naïve G/GEJ cancer: number analyzed (Participants) | 0 | 31
  Anti-PD-1/PD-L1 naïve G/GEJ cancer |  | 71.0 [52.0 to 85.8]

5. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS is defined as the time from the date of first dose to the date of first documentation of progressive disease assessed by the investigator per RECIST v1.1 or death, whichever occurs first. Safety analysis set is presented by indication group, as prespecified in the statistical analysis plan.
Time Frame: Up to approximately 4 years and 1 month
Population: The Safety Analysis Set includes all participants who received ≥ 1 dose of any study drug
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Sitravatinib Monotherapy | Sitravatinib + Tislelizumab
Number analyzed (Participants) | 24 | 83
Months
  Anti-PD-1/PD-L1 naïve or R/R HCC: number analyzed (Participants) | 24 | 0
  Anti-PD-1/PD-L1 naïve or R/R HCC | 6.8 [4.0 to 7.4] |
  Anti-PD-1/PD-L1 naïve HCC: number analyzed (Participants) | 0 | 27
  Anti-PD-1/PD-L1 naïve HCC |  | 6.8 [2.8 to 8.3]
  Anti-PD-1/PD-L1 R/R HCC: number analyzed (Participants) | 0 | 24
  Anti-PD-1/PD-L1 R/R HCC |  | 4.2 [2.7 to 6.8]
  Anti-PD-1/PD-L1 naïve G/GEJ cancer: number analyzed (Participants) | 0 | 32
  Anti-PD-1/PD-L1 naïve G/GEJ cancer |  | 3.6 [2.8 to 4.7]

6. Secondary Outcome: Maximum Plasma Concentration (Cmax) for Sitravatinib
Time Frame: Predose and up to 24 hours postdose on Cycle 1 Day 1 (C1D1) and Cycle 1 Day 21 (C1D21) (21 days in each cycle)
Population: The Sitravatinib Pharmacokinetic (PK) Analysis Set includes all participants who contributed ≥ 1 quantifiable PK sample for sitravatinib
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms/milliliter (ng/mL)
Arm/Group | Sitravatinib Monotherapy: 80 mg | Sitravatinib Monotherapy: 120 mg | Sitravatinib 80 mg + Tislelizumab | Sitravatinib 120 mg + Tislelizumab
Number analyzed (Participants) | 3 | 4 | 3 | 13
nanograms/milliliter (ng/mL)
  C1D1 | 27.11 (38.968) | 45.47 (67.213) | 37.02 (94.990) | 51.07 (52.218)
  C1D21: number analyzed (Participants) | 3 | 2 | 3 | 9
  C1D21 | 63.98 (3.060) | 69.30 (78.298) | 56.01 (103.431) | 62.38 (54.927)

7. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax) for Sitravatinib
Time Frame: Predose and up to 24 hours postdose on C1D1 and C1D21 (21 days in each cycle)
Population: The Sitravatinib PK Analysis Set includes all participants who contributed ≥ 1 quantifiable PK sample for sitravatinib
Measure: Median (Full Range); unit: Hours (h)
Arm/Group | Sitravatinib Monotherapy: 80 mg | Sitravatinib Monotherapy: 120 mg | Sitravatinib 80 mg + Tislelizumab | Sitravatinib 120 mg + Tislelizumab
Number analyzed (Participants) | 3 | 4 | 3 | 13
Hours (h)
  C1D1 | 10.0 [6.0 to 10.0] | 7.04 [4.0 to 10.0] | 10.0 [6.0 to 10.0] | 7.58 [1.8 to 12.4]
  C1D21: number analyzed (Participants) | 3 | 2 | 3 | 9
  C1D21 | 6.00 [6.0 to 12.0] | 3.04 [2.0 to 4.1] | 6.00 [0.5 to 10.0] | 9.15 [0.0 to 12.4]

8. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to the Last Measurable Time Point (AUC(0-t)) for Sitravatinib
Time Frame: Predose and up to 24 hours postdose on C1D1 and C1D21 (21 days in each cycle)
Population: The Sitravatinib PK Analysis Set includes all participants who contributed ≥ 1 quantifiable PK sample for sitravatinib
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Sitravatinib Monotherapy: 80 mg | Sitravatinib Monotherapy: 120 mg | Sitravatinib 80 mg + Tislelizumab | Sitravatinib 120 mg + Tislelizumab
Number analyzed (Participants) | 3 | 4 | 3 | 13
h*ng/mL
  C1D1 | 397.95 (25.561) | 761.95 (62.680) | 604.63 (118.143) | 840.74 (59.869)
  C1D21: number analyzed (Participants) | 3 | 2 | 3 | 9
  C1D21 | 1276.52 (3.498) | 1364.56 (116.841) | 1095.90 (119.358) | 1089.57 (91.752)

9. Secondary Outcome: Clearance After Oral Administration (CL/F) for Sitravatinib
Time Frame: Predose and up to 24 hours postdose on C1D1 and C1D21 (21 days in each cycle)
Population: The Sitravatinib PK Analysis Set includes all participants who contributed ≥ 1 quantifiable PK sample for sitravatinib
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters/hour
Arm/Group | Sitravatinib Monotherapy: 80 mg | Sitravatinib Monotherapy: 120 mg | Sitravatinib 80 mg + Tislelizumab | Sitravatinib 120 mg + Tislelizumab
Number analyzed (Participants) | 3 | 1 | 1 | 6
Liters/hour
  C1D1: number analyzed (Participants) | 1 | 1 | 0 | 5
  C1D1 | 92.58 (NA) — NA = not estimable due to single participant | 35.23 (NA) — NA = not estimable due to single participant |  | 82.77 (62.096)
  C1D21: number analyzed (Participants) | 3 | 0 | 1 | 6
  C1D21 | 63.76 (5.016) |  | 29.14 (NA) — NA = not estimable due to single participant | 78.31 (44.296)

10. Secondary Outcome: Area Under the Plasma Concentration-time Curve During the Dosing Interval (AUC(0-tau)) for Sitravatinib
Time Frame: Predose and up to 24 hours postdose on C1D1 and C1D21 (21 days in each cycle)
Population: The Sitravatinib PK Analysis Set includes all participants who contributed ≥ 1 quantifiable PK sample for sitravatinib
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Sitravatinib Monotherapy: 80 mg | Sitravatinib Monotherapy: 120 mg | Sitravatinib 80 mg + Tislelizumab | Sitravatinib 120 mg + Tislelizumab
Number analyzed (Participants) | 3 | 2 | 1 | 6
h*ng/mL
  C1D1: number analyzed (Participants) | 1 | 2 | 0 | 6
  C1D1 | 535.82 (NA) — NA = not estimable due to single participant | 686.11 (122.918) |  | 639.49 (63.908)
  C1D21: number analyzed (Participants) | 3 | 0 | 1 | 6
  C1D21 | 1254.71 (5.016) |  | 2745.23 (NA) — NA = not estimable due to single participant | 1532.33 (44.296)

11. Secondary Outcome: Observed Accumulation Ratio (Ro) for AUC(0-tau) for Sitravatinib
Time Frame: Predose and up to 24 hours postdose on C1D1 and C1D21 (21 days in each cycle)
Population: The Sitravatinib PK Analysis Set includes all participants who contributed ≥ 1 quantifiable PK sample for sitravatinib
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Sitravatinib Monotherapy: 80 mg | Sitravatinib Monotherapy: 120 mg | Sitravatinib 80 mg + Tislelizumab | Sitravatinib 120 mg + Tislelizumab
Number analyzed (Participants) | 1 | 0 | 0 | 2
Ratio | NA [NA to NA] — NA = not estimable due to low number of participants with events |  |  | 3.94 [0.09 to 165.95]

12. Secondary Outcome: Observed Accumulation Ratio (Ro) for Cmax for Sitravatinib
Time Frame: Predose and up to 24 hours postdose on C1D1 and C1D21 (21 days in each cycle)
Population: The Sitravatinib PK Analysis Set includes all participants who contributed ≥ 1 quantifiable PK sample for sitravatinib
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Sitravatinib Monotherapy: 80 mg | Sitravatinib Monotherapy: 120 mg | Sitravatinib 80 mg + Tislelizumab | Sitravatinib 120 mg + Tislelizumab
Number analyzed (Participants) | 3 | 2 | 3 | 8
Ratio | 2.36 [0.99 to 5.63] | 2.12 [0.72 to 6.25] | 1.51 [0.92 to 2.48] | 1.48 [0.89 to 2.47]

13. Secondary Outcome: Plasma Concentrations of Sitravatinib
Time Frame: Predose and 6 hours postdose in Cycle 5 Day 1 (21 days in each cycle)
Population: The Sitravatinib PK Analysis Set includes all participants who contributed ≥ 1 quantifiable PK sample for sitravatinib
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Sitravatinib Monotherapy: Sitravatinib 80 mg or 120 mg orally once daily in 21-day cycles in participants with unresectable locally advanced or metastatic HCC
Arm/Group | Sitravatinib Monotherapy | Sitravatinib + Tislelizumab
Number analyzed (Participants) | 5 | 19
ng/mL
  Predose: Anti-PD-1/PD-L1 naïve or R/R HCC: number analyzed (Participants) | 5 | 0
  Predose: Anti-PD-1/PD-L1 naïve or R/R HCC | 31.64 (18.492) |
  Postdose: Anti-PD-1/PD-L1 naïve or R/R HCC: number analyzed (Participants) | 5 | 0
  Postdose: Anti-PD-1/PD-L1 naïve or R/R HCC | 48.12 (34.581) |
  Predose: Anti-PD-1/PD-L1 naïve HCC: number analyzed (Participants) | 0 | 5
  Predose: Anti-PD-1/PD-L1 naïve HCC |  | 23.54 (1435.332)
  Postdose: Anti-PD-1/PD-L1 naïve HCC: number analyzed (Participants) | 0 | 5
  Postdose: Anti-PD-1/PD-L1 naïve HCC |  | 77.40 (65.582)
  Predose: Anti-PD-1/PD-L1 R/R HCC: number analyzed (Participants) | 0 | 8
  Predose: Anti-PD-1/PD-L1 R/R HCC |  | 35.95 (91.411)
  Postdose: Anti-PD-1/PD-L1 R/R HCC: number analyzed (Participants) | 0 | 8
  Postdose: Anti-PD-1/PD-L1 R/R HCC |  | 54.05 (49.017)
  Predose: Anti-PD-1/PD-L1 naïve G/GEJ cancer: number analyzed (Participants) | 0 | 6
  Predose: Anti-PD-1/PD-L1 naïve G/GEJ cancer |  | 31.13 (66.433)
  Postdose: Anti-PD-1/PD-L1 naïve G/GEJ cancer: number analyzed (Participants) | 0 | 6
  Postdose: Anti-PD-1/PD-L1 naïve G/GEJ cancer |  | 42.22 (32.131)

ADVERSE EVENTS:
Time Frame: From first dose up to 30 days after last dose of study drug(s) or initiation of new anticancer therapy; up to approximately 4 years and 1 month
Groups:
- Sitravatinib 120 mg + Tislelizumab: Sitravatinib 120 mg orally once daily in 21-day cycles with tislelizumab 200 mg intravenously (IV) once every 3 weeks in participants with unresectable locally advanced or metastatic HCC or G/GEJ cancer
Arm/Group | Sitravatinib Monotherapy: 80 mg | Sitravatinib Monotherapy: 120 mg | Sitravatinib 80 mg + Tislelizumab | Sitravatinib 120 mg + Tislelizumab
All-Cause Mortality (participants affected / at risk) | 0/3 | 12/24 | 2/3 | 53/81
Serious Adverse Events (participants affected / at risk) | 1/3 | 7/24 | 2/3 | 31/81
Other Adverse Events (participants affected / at risk) | 3/3 | 24/24 | 3/3 | 78/81
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sitravatinib Monotherapy: 80 mg (N=3) | Sitravatinib Monotherapy: 120 mg (N=24) | Sitravatinib 80 mg + Tislelizumab (N=3) | Sitravatinib 120 mg + Tislelizumab (N=81)
Hypersplenism (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Death (General disorders) | 0 (0) | 0 (0) | 1 (1) | 7 (7)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Jaundice cholestatic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tuberculosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myocardial necrosis marker increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatic encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Immune-mediated encephalitis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Loss of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nephrotic syndrome (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Venous thrombosis limb (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sitravatinib Monotherapy: 80 mg (N=3) | Sitravatinib Monotherapy: 120 mg (N=24) | Sitravatinib 80 mg + Tislelizumab (N=3) | Sitravatinib 120 mg + Tislelizumab (N=81)
Anaemia (Blood and lymphatic system disorders) | 1 (2) | 5 (9) | 1 (1) | 22 (35)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypersplenism (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Splenomegaly (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (3)
Extrasystoles (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Supraventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (3)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Deafness (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 7 (7)
Hypothyroidism (Endocrine disorders) | 2 (2) | 3 (3) | 1 (1) | 16 (16)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 4 (4) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 4 (4) | 0 (0) | 1 (5)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 13 (15)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 14 (27) | 0 (0) | 27 (51)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Duodenitis (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 3 (3) | 1 (1) | 10 (12)
Oral pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Retching (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Toothache (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (3) | 0 (0) | 1 (1) | 13 (14)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 7 (9)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Fatigue (General disorders) | 0 (0) | 1 (2) | 1 (1) | 9 (9)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Malaise (General disorders) | 0 (0) | 1 (1) | 0 (0) | 4 (4)
Peripheral swelling (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 7 (8)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 3 (3) | 0 (0) | 3 (5)
Hepatic pain (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Portal hypertension (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Alanine aminotransferase increased (Investigations) | 2 (4) | 13 (23) | 3 (4) | 41 (71)
Alpha hydroxybutyrate dehydrogenase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 9 (25)
Aspartate aminotransferase increased (Investigations) | 2 (4) | 13 (22) | 3 (6) | 41 (78)
Bilirubin conjugated increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 6 (9)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 3 (4) | 0 (0) | 15 (21)
Blood bilirubin increased (Investigations) | 1 (1) | 3 (4) | 0 (0) | 19 (29)
Blood bilirubin unconjugated increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Blood creatine phosphokinase MB increased (Investigations) | 0 (0) | 2 (2) | 1 (1) | 25 (55)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 1 (3) | 0 (0) | 15 (36)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 5 (5)
Blood fibrinogen increased (Investigations) | 0 (0) | 1 (3) | 0 (0) | 2 (6)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 3 (3) | 0 (0) | 12 (27)
Blood pressure increased (Investigations) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Blood thyroid stimulating hormone increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 14 (18)
C-reactive protein increased (Investigations) | 0 (0) | 2 (3) | 0 (0) | 3 (11)
Fibrin D dimer increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 3 (7)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 5 (7) | 0 (0) | 14 (25)
Myocardial necrosis marker increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (3) | 2 (3) | 0 (0) | 5 (12)
Neutrophil count increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Platelet count decreased (Investigations) | 2 (3) | 10 (13) | 0 (0) | 22 (40)
Thyroglobulin decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thyroxine free decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 5 (6)
Urinary occult blood positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 5 (10)
Weight decreased (Investigations) | 3 (3) | 6 (7) | 1 (1) | 14 (17)
White blood cell count decreased (Investigations) | 1 (4) | 4 (5) | 0 (0) | 14 (31)
White blood cell count increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 3 (3) | 1 (1) | 17 (18)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 7 (7)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (4) | 0 (0) | 6 (10)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 3 (5) | 2 (2) | 34 (44)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 4 (4)
Hypochloraemia (Metabolism and nutrition disorders) | 0 (0) | 2 (3) | 0 (0) | 8 (9)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (5) | 5 (7) | 1 (1) | 9 (22)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 4 (4)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (2) | 2 (3) | 2 (2) | 10 (11)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 5 (6)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 7 (9)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Vertebral artery occlusion (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vertebral artery stenosis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (4)
Nephrotic syndrome (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 2 (2) | 13 (24) | 2 (2) | 44 (69)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 4 (4)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (7) | 0 (0) | 8 (10)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 5 (5)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 2 (2) | 17 (20) | 0 (0) | 31 (32)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (4) | 0 (0) | 7 (8)
Skin disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aortic thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 3 (3) | 4 (11) | 2 (3) | 28 (32)
Venous thrombosis limb (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
BeiGene has 18 months from the end of the study at all sites to publish overall study results. After the 1st multi-site publication or the expiration of publication period, Investigators are free to publish/present the results of the study. Investigators must submit all draft publications/presentations to us for review 60 days prior to the planned publication/presentation date. BeiGene may request deletion of its confidential information & may request a further delay to protect its IP rights.

DOCUMENTS (2):
  • Study Protocol (2020-04-28): https://cdn.clinicaltrials.gov/large-docs/73/NCT03941873/Prot_000.pdf
  • Statistical Analysis Plan (2023-04-10): https://cdn.clinicaltrials.gov/large-docs/73/NCT03941873/SAP_001.pdf